CLINICAL TRIAL: NCT03389802
Title: Phase I Study to Evaluate the Safety and Tolerability of the CD40 Agonistic Monoclonal Antibody APX005M in Pediatric Subjects With Recurrent/Refractory Brain Tumors and Newly Diagnosed Brain Stem Glioma
Brief Title: Phase I Study of APX005M in Pediatric Central Nervous System Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: American Lebanese Syrian Associated Charities (Other); Pyxis Oncology, Inc (Industry); Solving Kids' Cancer (Other); Ty Louis Campbell Foundation (Other); A Kids' Brain Tumor Cure Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-051; UM1CA081457 (NIH); PBTC-051 (Other: Pediatric Brain Tumor Consortium); PBTC-051 (Other: CTEP); NCI-2017-01235 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-12-15; First posted 2018-01-04 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma Multiforme; High-grade Astrocytoma Not Otherwise Specified (NOS); CNS Primary Tumor, Not Otherwise Specified (NOS); Ependymoma, Not Otherwise Specified (NOS); Diffuse Intrinsic Pontine Gliomas (DIPG); Medulloblastoma
MeSH Terms: conditions — Glioblastoma; Ependymoma; Medulloblastoma

STUDY DESIGN:
Intervention Model Description: Stratum 1: Recurrent or refractory primary malignant CNS tumor patients; Stratum 2: Newly diagnosed DIPG patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stratum 1 (Experimental): The recurrent, progressive, or refractory primary malignant non-brainstem CNS tumor patients will be treated with APX005M.
  Interventions: Biological: APX005M treatment for recurrent or refractory primary malignant CNS tumor patients
- Stratum 2 (Experimental): The newly diagnosed diffuse intrinsic pontine gliomas (DIPGs) patients will be treated with APX005M.
  Interventions: Biological: APX005M treatment for newly diagnosed DIPG patients

INTERVENTIONS:
Biological: APX005M treatment for recurrent or refractory primary malignant CNS tumor patients — APX005M dosing will begin at 0.1 mg/kg, the APX005M dose may be increased (0.3, 0.45, 0.6 mg/kg) or decreased (0.03 mg/kg) in subsequent cohorts until the maximum tolerated dose (MTD) is reached or until dose level 3 (0.6 mg/kg) is complete without the MTD being defined.
  APX005M will be administered at the assigned dose level every 21 days (3 weeks). Patients may continue to receive APX005M for 36 courses (approximately 2 years) or until disease progression, unacceptable toxicity or death, whichever occurs first.
  Arms: Stratum 1
Biological: APX005M treatment for newly diagnosed DIPG patients — The starting dose of APX005M for the DIPG patients will be one dose level below the recommended phase II dose (RP2D) determined in Stratum 1 patients. The dose may be decreased or increased to the RP2D established in Stratum 1.
  APX005M will be administered at the assigned dose level every 21 days (3 weeks). Patients may continue to receive APX005M for 36 courses (approximately 2 years) or until disease progression, unacceptable toxicity or death, whichever occurs first.
  Arms: Stratum 2

SUMMARY:
This phase I trial studies the side effects and best dose of APX005M in treating younger patients with primary malignant central nervous system tumor that is growing, spreading, or getting worse (progressive), or newly diagnosed diffuse intrinsic pontine glioma. APX005M can trigger activation of B cells, monocytes, and dendritic cells and stimulate cytokine release from lymphocytes and monocytes. APX005M can mediate a direct cytotoxic effect on CD40+ tumor cells.

DETAILED DESCRIPTION:
This is a multicenter phase I trial of APX005M in patients with recurrent or refractory primary malignant central nervous system tumor, or newly diagnosed diffuse intrinsic pontine glioma.

APX005M is a humanized IgG1κ mAb that binds to CD40. APX005M binds to both human and cynomolgus monkey CD40 with high affinity, triggering activation of B cells, monocytes, and dendritic cells and stimulating cytokine release from both human and monkey lymphocytes and monocytes. APX005M does not bind to mouse or rat CD40. CD40 is also expressed on many human tumor cells, and APX005M can mediate a direct cytotoxic effect on CD40+ tumor cells.

Activation of CD40 on tumor cells results in tumor cell apoptosis and inhibition of tumor growth. CD40 agonistic antibodies have demonstrated potent antitumor immune response stimulation in both animal models and cancer patients. Due to its action on both immune and tumor cells, CD40 has been studied as a target for novel cancer immunotherapy.

Apexigen has declared the adult recommended phase 2 dose to be 0.3 mg/kg because no dose limiting toxicities were encountered at that dose and the pharmacodynamic profile was similar to the 1 mg/kg maximally tolerated dose. This phase 1 clinical trial is to study APX005M in children with central nervous system tumors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis -- Stratum 1: Recurrent or refractory primary malignant CNS tumor patients Patients with a histologically confirmed diagnosis of a primary malignant non-brainstem CNS tumor (excluding DIPG patients) that is recurrent, progressive, or refractory. All tumors must have histologic verification at either the time of diagnosis or recurrence except patients with marker (+) CNS germ cell tumors.

Stratum 2: Newly diagnosed DIPG patients (on-hold until pediatric RP2D has been established in Stratum 1) Patients with diffuse intrinsic pontine gliomas (DIPGs) will be eligible 6 to 14 weeks post-completion of radiation therapy if they do not have any evidence of progression. Patients with newly diagnosed DIPGs, defined as tumors with a pontine epicenter and diffuse involvement of 2/3 or more of the pons, are eligible without histologic confirmation. Patients with pontine tumors that do not meet these criteria or not considered to be typical intrinsic pontine gliomas will only be eligible if the tumors have been biopsied and (1) are proven to be an anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, anaplastic mixed glioma or fibrillary astrocytoma or (2) have a histone mutation typically seen in DIPG. Patients with disseminated disease are not eligible, and MRI of spine must be performed if disseminated disease is suspected by the treating physician.

* Available Pre-trial Tumor Tissue -- Stratum 1: Recurrent or refractory primary malignant CNS tumor patients must have adequate pre-trial frozen or FFPE tumor material (minimum of 10 unstained slides) available for use in the tumor mutation burden studies (section 9.1.5).

Stratum 2: Patients with DIPG who have pre-trial tumor tissue available are requested to submit tissue; however, this is not required for eligibility.

* Age -- Patient must be ≥ 1 and ≤ 21 years of age at the time of enrollment.
* Prior Therapy -- Newly Diagnosed DIPG patients Patients must have not received any prior therapy for treatment of their current CNS malignancy other than radiation therapy.

Refractory/Recurrent patients Patients must have recovered from the acute treatment related toxicities (defined as < grade 1) of all prior chemotherapy, immunotherapy, radiotherapy or any other treatment modality prior to entering this study.

Myelosuppressive chemotherapy -- Patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days if nitrosourea.

Biological agent: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the biologic agent ≥ 7 days prior to study enrollment.

For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.

Monoclonal antibody treatment and agents with known prolonged half-lives: At least three half-lives must have elapsed prior to enrollment.

Radiation --

Patients must have had their last fraction of:

Craniospinal irradiation (>24Gy) or total body irradiation or radiation to greater than 50% of pelvis > 3 months prior to enrollment.

Focal irradiation >6 weeks prior to enrollment Local palliative irradiation (small port) ≥4 weeks

Autologous Stem Cell Transplant -- Patient must be ≥ 6 months since autologous bone marrow/stem cell transplant prior to enrollment and have CD4 counts above 200/mm3.

Surgery -- Patients must be at least 4 weeks (28 days) from major surgery and fully recovered from all acute effects of prior surgical intervention.

* Inclusion of Women and Minorities -- Both males and females of all races and ethnic groups are eligible for this study
* Neurologic Status -- Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment.

Patients with seizure disorders may be enrolled if seizures are well controlled.

• Performance Status -- Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) assessed within two weeks of enrollment must be ≥ 60. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

• Organ Function --

Patients must have adequate organ and bone marrow function as defined below:

Absolute Neutrophil Count (ANC) ≥ 1.0 x 109 cells/ L Platelets ≥ 100 x 109 cells/L (unsupported, defined as no platelet transfusion within 7 days) Hemoglobin ≥ 8 g/dL (may receive transfusions) Total bilirubin ≤1.5 times institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤ 3 x institutional upper limit of normal (ULN) Albumin ≥ 3 g/dl Serum creatinine based on age/gender as noted below. Patients that do not meet the criteria below but have a 24 hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 mL/min/1.73 m2 are eligible.

Age Maximum Serum Creatinine (mg/dL) 1 to < 2 years 0.6, 0.6 (M, F); 2 to < 6 years 0.8, 0.8 (M, F); 6 to < 10 years 1, 1 (M, F); 10 to < 13 years 1.2, 1.2 (M, F); 13 to < 16 years 1.5, 1.4 (M, F); ≥ 16 years 1.7, 1.4 (M, F).

• Cardiac Function: Left Ventricular Ejection Fraction (LVEF) > 50% ECG QTc ≤ 450 msec

• Pulmonary Function: Oxygen saturation as measured by pulse oximetry is > 93% on room air and no evidence of dyspnea at rest

• Growth Factors -- Patients must be off all colony- forming growth factor(s) for at least 1 week prior to enrollment (i.e., filgrastim, sargramostim or erythropoietin). 2 weeks must have elapsed if patients received PEG formulations.

* Pregnancy Status -- Female patients of childbearing potential must have a negative serum or urine pregnancy test.
* Pregnancy Prevention -- Female subjects with childbearing potential and male subjects should use effective contraception methods (or abstain from sexual activity) while being treated with APX005M and for 30 days following treatment.
* Informed Consent -- The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines.

Exclusion Criteria:

• Concurrent Illness -- Patients with any clinically significant unrelated systemic illness (serious infections Grade ≥ 2 or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.

Patients with a history of any other malignancy, except patients with a secondary brain tumor if the patient's first malignancy has been in remission for at least 5 years from the end of treatment.

• Concurrent Therapy -- Patients who are receiving any other anticancer or investigational drug therapy.

Patients requiring systemic treatment with either corticosteroids (greater than physiologic replacement, defined as dexamethasone 0.75 mg/m2/day) or other immunosuppressive medications within 14 days of study drug administration will be excluded. However, patients who require intermittent use of bronchodilators or local steroid injections will not be excluded from the study. Please see section 5.3 for a list of acceptable and unacceptable concomitant medications as well as reporting requirements.

• Presence of Bulky Tumor --

Patients with bulky tumor on imaging are ineligible. Bulky tumor is defined as:

Tumor with any evidence of uncal herniation or midline shift Tumor that in the opinion of the site investigator, shows significant mass effect

* Allergy -- Patients with a history of severe (Grade ≥ 3) hypersensitivity reaction to a monoclonal antibody are ineligible.
* Allogeneic Hematopoietic Stem Cell Transplantation -- Patients who have received allogeneic hematopoietic stem cell transplantation are ineligible.
* Autoimmune Diseases -- Patients with active autoimmune disease or documented history of autoimmune disease/syndrome that requires ongoing systemic steroids or systemic immunosuppressive agents, except Patients with vitiligo or well controlled asthma/atopy Patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome
* Inability to Participate -- Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions.
* Bleeding Disorder -- Patients with a known coagulopathy or bleeding diathesis or require the use of systemic anticoagulant medication are not eligible.
* Pregnancy Status -- Female patients must not be pregnant or breast-feeding.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-11-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Dunkel, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Childrens Hospital-Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children Hospital Medical Center, Cincinnati, Ohio
  - Children Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients ≥1 and ≤21 years of age with recurrent or refractory primary malignant central nervous system (CNS) tumors (Stratum 1) or newly diagnosed diffuse intrinsic pontine glioma (DIPG) (Stratum 2) were enrolled at Pediatric Brain Tumor Consortium (PBTC) member institutions. The first patient was enrolled on 3/1/2018 and the last patient was enrolled on 1/20/2023. Accrual was closed after the maximum tolerated dose/recommended phase II dose was determined for both strata.
Pre-assignment Details: Patients with recurrent or refractory primary malignant CNS tumors were enrolled on stratum 1, and patients with newly diagnosed diffuse intrinsic pontine glioma (DIPG) were enrolled on stratum 2. A total of 32 patients were enrolled (31 eligible). Twenty-one (21) stratum 1 patients were enrolled; 1 of these patients was deemed to be ineligible as an eligibility assessment was not performed. Eleven (11) stratum 2 patients were enrolled (all deemed eligible).
Groups:
- Stratum 1, Dose Level 1: Patients with recurrent or refractory primary malignant CNS tumors received APX005M on day 1 of each 21-day course at 0.1 mg/kg for up to 36 courses or until disease progression, unacceptable toxicity, or death.
- Stratum 1, Dose Level 2: Patients with recurrent or refractory primary malignant CNS tumors received APX005M on day 1 of each 21-day course at 0.3 mg/kg for up to 36 courses or until disease progression, unacceptable toxicity, or death.
- Stratum 1, Dose Level 3: Patients with recurrent or refractory primary malignant CNS tumors received APX005M on day 1 of each 21-day course at 0.6 mg/kg for up to 36 courses or until disease progression, unacceptable toxicity, or death.
- Stratum 2, Dose Level 2: Patients with newly diagnosed diffuse intrinsic pontine glioma (DIPG) received APX005M on day 1 of each 21-day course at 0.3 mg/kg for up to 36 courses or until disease progression, unacceptable toxicity, or death.
- Stratum 2, Dose Level 3: Patients with newly diagnosed diffuse intrinsic pontine glioma (DIPG) received APX005M on day 1 of each 21-day course at 0.6 mg/kg for up to 36 courses or until disease progression, unacceptable toxicity, or death.
Period: Overall Study
Arm/Group | Stratum 1, Dose Level 1 | Stratum 1, Dose Level 2 | Stratum 1, Dose Level 3 | Stratum 2, Dose Level 2 | Stratum 2, Dose Level 3
Started | 3 | 3 | 15 | 6 | 5
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 15 | 6 | 5
Not completed — Lack of Efficacy | 3 | 3 | 13 | 6 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 4
Not completed — Subject deemed ineligible after enrollment | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The one stratum 1, dose level 3 participant found to be ineligible after enrollment was excluded. Summary statistics for baseline characteristics are shown for eligible patients only (n=31).
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1, Dose Level 1 | Stratum 1, Dose Level 2 | Stratum 1, Dose Level 3 | Stratum 2, Dose Level 2 | Stratum 2, Dose Level 3 | Total
Number analyzed (Participants) | 3 | 3 | 14 | 6 | 5 | 31
Age, Continuous [Median (Full Range); unit: Year] — The median and full range for age at the time of study enrollment was reported (in years).
  Year | 4.2 [3.4 to 14.6] | 13.2 [8.9 to 21.9] | 9.7 [2.2 to 20.6] | 6.6 [1.4 to 10.4] | 8.8 [2.8 to 10.6] | 8.9 [1.4 to 21.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 7 | 4 | 5 | 18
  Male | 2 | 2 | 7 | 2 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 4 | 3 | 2 | 11
  Not Hispanic or Latino | 2 | 1 | 9 | 3 | 2 | 17
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 2
  White | 2 | 3 | 10 | 4 | 0 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced Dose-limiting Toxicities (DLTs)
Description: DLTs were defined as adverse events (AE) at least possibly attributed to APX005M that occurred during the first 2 courses (6 weeks) following APX005M administration. DLTs included any APX005M-related AE that led to dose reduction or permanent cessation of therapy or resulted in a treatment delay >2 weeks. Hematologic DLTs included grade 3 neutropenia with fever, any grade 4 hematologic toxicity except lymphopenia, and grade 3 thrombocytopenia on 2 separate days or requiring platelet transfusion on 2 days within a 7-day period. Non-hematologic DLTs included any grade 4 non-hematologic toxicity, grade 3 or higher cytokine release syndrome, or any grade 3 non-hematologic toxicity with some exceptions such as grade 3 nausea/vomiting <5 days or grade 3 diarrhea that responded to treatment within 5 days.
Time Frame: 6 weeks
Population: Patients who were evaluable for DLT assessment were included in this analysis. Of 31 eligible patients enrolled, 2 patients were not evaluable for DLT assessment due to early disease progression (received less than 2 doses of therapy).
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1, Dose Level 1 | Stratum 1, Dose Level 2 | Stratum 1, Dose Level 3 | Stratum 2, Dose Level 2 | Stratum 2, Dose Level 3
Number analyzed (Participants) | 3 | 3 | 12 | 6 | 5
Participants | 0 | 0 | 2 | 0 | 3

2. Primary Outcome: Maximum Tolerated Dose (MTD) and/or Recommended Phase II Dose (RP2D) of APX005M in Stratum 1
Description: Based on the 3+3 design, the MTD of APX005M was empirically defined as the highest dose level at which six patients were treated with at most one patient experiencing a DLT, and the next higher dose level was determined to be too toxic. A total of 12 subjects were to be treated at the MTD/RP2D to further define the toxicity profile. Stratum 1 consisted of patients with recurrent or refractory primary malignant central nervous system tumors.
Time Frame: 6 weeks (first 2 courses of treatment)
Population: Patients who were enrolled on Stratum 1 and evaluable for dose-finding assessment were used to determine the MTD for Stratum 1. Of 20 eligible patients enrolled on Stratum 1, 2 were not evaluable for dose-finding assessment due to early progressive disease (these 2 participants received less than 2 doses of treatment). The remaining 18 patients were used to determine the MTD/RP2D for Stratum 1.
Measure: Number; unit: mg/kg
Groups:
- Stratum 1: Recurrent, progressive, or refractory primary malignant non-brainstem CNS tumor patients treated with APX005M.
  The dose levels studied were 0.1 mg/kg (dose level 1), 0.3 mg/kg (dose level 2), and 0.6 mg/kg (dose level 3).
  APX005M was administered at the assigned dose level every 21 days (3 weeks). Patients could receive APX005M for 36 courses (approximately 2 years) or until disease progression, unacceptable toxicity or death.
Arm/Group | Stratum 1
Number analyzed (Participants) | 18
mg/kg | 0.6

3. Primary Outcome: Maximum Tolerated Dose (MTD) and/or Recommended Phase II Dose (RP2D) of APX005M in Stratum 2
Description: The starting dose level for Stratum 2 was one dose level below the RP2D determined in Stratum 1. If there were no dose-limiting toxicities in the first 3 patients enrolled on Stratum 2, then we escalated to the Stratum 1 RP2D and could treat 6 diffuse intrinsic pontine glioma (DIPG) patients simultaneously. The RP2D was defined as the dose level at which 6 patients were treated with no more than one dose-limiting toxicity. Stratum 2 patients were those with newly diagnosed diffuse intrinsic pontine glioma (DIPG).
Time Frame: 6 weeks (first 2 courses of treatment)
Population: Patients who were enrolled on Stratum 2 and were evaluable for dose-finding assessment were used to determine the MTD for Stratum 2. Of 11 patients enrolled on Stratum 2, all were evaluable for dose-finding assessment and used to determine the MTD for Stratum 2.
Measure: Number; unit: mg/kg
Groups:
- Stratum 2: Newly diagnosed diffuse intrinsic pontine gliomas (DIPGs) patients treated with APX005M.
  The dose levels studied were 0.3 mg/kg (dose level 2) and 0.6 mg/kg (dose level 3). Dose level 2 was selected as the starting dose level for Stratum 2 as it was one dose level lower than the Stratum 1 MTD/RP2D.
  APX005M was administered at the assigned dose level every 21 days (3 weeks). Patients could receive APX005M for 36 courses (approximately 2 years) or until disease progression, unacceptable toxicity or death.
Arm/Group | Stratum 2
Number analyzed (Participants) | 11
mg/kg | 0.3

4. Primary Outcome: Serum Concentration of APX005M
Description: Serial blood samples for APX005M pharmacokinetic studies were collected during courses 1 and 2 at pre-dose, at the end of infusion, and at 4, 24 ± 1 (Day 2), and 168 ± 4 hours (Day 8) from the start of infusion in that course and during courses 3 and 4 at pre-dose and end of induction.
Time Frame: 12 weeks
Reporting Status: Not Posted, anticipated posting 2025-09

5. Secondary Outcome: Overall Survival for Stratum 2 (DIPG) Patients
Description: Overall survival was defined as the time interval from treatment initiation to death from any cause or to date of last follow-up for survivors. Survival was estimated using the method of Kaplan and Meier. The 1-year estimate of survival is reported with a 95% confidence interval; estimates are reported by dose level. Stratum 2 patients were those with newly diagnosed diffuse intrinsic pontine glioma (DIPG).
Time Frame: 1 year
Population: Newly diagnosed DIPG patients who were enrolled on Stratum 2 and received at least one dose of APX005M were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Stratum 2, Dose Level 2 | Stratum 2, Dose Level 3
Number analyzed (Participants) | 6 | 5
Percent probability | 40.0 [4.9 to 75.1] | 25.0 [0.0 to 55.0]

6. Secondary Outcome: Progression-free Survival for Stratum 2 (DIPG) Patients
Description: Progression-free survival (PFS) was defined as the time interval from treatment initiation to date of first event (relapsed or progressive disease based on imaging or clinical progression or death from any cause) or to the date of last follow-up for patients without events. PFS was estimated using the method of Kaplan and Meier. The 1-year estimate of PFS is reported with a 95% confidence interval. PFS estimates were reported separately by dose level. Stratum 2 patients were those with newly diagnosed diffuse intrinsic pontine glioma (DIPG).
Time Frame: 1 year
Population: Newly diagnosed DIPG patients who were enrolled on Stratum 2 and received at least one dose of APX005M are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Stratum 2, Dose Level 2 | Stratum 2, Dose Level 3
Number analyzed (Participants) | 6 | 5
Percent probability | 16.7 [0.0 to 37.9] | 26.7 [0.0 to 58.3]

7. Secondary Outcome: Overall Response Rate for Stratum 2 (DIPG) Patients
Description: Complete or partial responses were considered responses. Response was evaluated by imaging or clinical progression. The response rate (percentage of participants with responses) is reported with a 95% Blyth-Still-Casella confidence interval. Response rates are reported separately by dose level.
Time Frame: Up to 2 years
Population: Stratum 2 patients with measurable disease present at baseline who received at least one dose of therapy and had their disease re-evaluated were considered evaluable for objective response. Two participants were considered not evaluable as they did not have their disease re-evaluated.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Stratum 2, Dose Level 2 | Stratum 2, Dose Level 3
Number analyzed (Participants) | 6 | 3
percentage | 0 [0.0 to 40.2] | 0 [0.0 to 63.2]

8. Secondary Outcome: Duration of Response for Stratum 2 (DIPG) Patients
Description: Complete or partial responses were considered responses. Response was evaluated by imaging or clinical progression. Duration of response was measured from the time measurement criteria are met for complete or partial response until the first date that recurrent or progressive disease was objectively documented.
Time Frame: Up to 2 years
Population: Of the 11 Stratum 2 patients (6 dose level 2, 5 dose level 3), 2 (both in dose level 3) were considered not evaluable for response. As no participants had complete or partial responses, it was not possible to calculate duration of response.
Arm/Group | Stratum 2, Dose Level 2 | Stratum 2, Dose Level 3
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Concentration of the Cytokine Tumor Necrosis Factor-alpha (TNF-alpha)
Description: Concentration of the cytokine Tumor Necrosis Factor-alpha (TNF-alpha) (in pg/ml)
Time Frame: Pre-treatment and up to 9 weeks post-treatment
Reporting Status: Not Posted, anticipated posting 2025-07

10. Other Pre Specified Outcome: Concentration of the Cytokine Interleukin-8 (IL-8)
Description: Concentration of the cytokine Interleukin-8 (IL-8) (in pg/ml)
Time Frame: Pre-treatment and up to 9 weeks post-treatment
Reporting Status: Not Posted, anticipated posting 2025-07

11. Other Pre Specified Outcome: T Cell Phenotypes in Human PBMC
Description: Characterization of T cell phenotypes in human PBMC
Time Frame: Pre-treatment and up to 9 weeks post-treatment
Reporting Status: Not Posted, anticipated posting 2025-07

12. Other Pre Specified Outcome: Mutational Burden Based on Whole Exome Sequencing of Tumor Tissue and PBMC
Description: Mutational burden as detected by comparing whole exome sequencing of tumor tissue and PBMC
Time Frame: Day 0 of treatment
Reporting Status: Not Posted, anticipated posting 2025-07

13. Other Pre Specified Outcome: Mutational Burden Based on RNAseq of Tumor Tissue and PBMC
Description: Mutation burden as detected by comparing the RNA sequencing of tumor tissue and PBMC
Time Frame: Day 0 of treatment
Reporting Status: Not Posted, anticipated posting 2025-07

14. Other Pre Specified Outcome: Mutational Burden Based on TCR Sequencing
Description: Mutational burden as detected by comparing the TCR sequencing of tumor tissue and/or PBMC. For Stratum 2 (DIPG) patients without tumor samples, TCRseq analysis will be performed, which only requires PBMCs.
Time Frame: Day 0 of treatment
Reporting Status: Not Posted, anticipated posting 2025-07

15. Other Pre Specified Outcome: Incidence of Anti-APX005M Antibodies
Description: Serial blood samples for anti-drug-antibodies (ADA) are to be collected prior to dosing on courses 1 through 4, then every third course (courses 7 and 10), and then every 4 courses (courses 14, 18, 22, 26, 30, 34) until the end of therapy visit and collected into serum tubes.
Time Frame: Approximately 2 years
Reporting Status: Not Posted, anticipated posting 2025-07

ADVERSE EVENTS:
Time Frame: Approximately 3 years after start of treatment
Description: Adverse events were graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. Per Section 7 of the protocol, all adverse events grades 3 through 4 and deaths, regardless of attribution to study drug, were collected, and adverse events grades 1 and 2 were to be recorded only if the attribution was at least possibly related to study drug. Of note, all deaths on this study were due to disease. All eligible patients are included in adverse event reporting.
Arm/Group | Stratum 1, Dose Level 1 | Stratum 1, Dose Level 2 | Stratum 1, Dose Level 3 | Stratum 2, Dose Level 2 | Stratum 2, Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 5/14 | 4/6 | 4/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 4/14 | 1/6 | 5/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 14/14 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1, Dose Level 1 (N=3) | Stratum 1, Dose Level 2 (N=3) | Stratum 1, Dose Level 3 (N=14) | Stratum 2, Dose Level 2 (N=6) | Stratum 2, Dose Level 3 (N=5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1, Dose Level 1 (N=3) | Stratum 1, Dose Level 2 (N=3) | Stratum 1, Dose Level 3 (N=14) | Stratum 2, Dose Level 2 (N=6) | Stratum 2, Dose Level 3 (N=5)
Lymphocyte count decreased (Investigations) | 2 (3) | 2 (6) | 7 (18) | 2 (6) | 4 (9)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 3 (7) | 9 (22) | 3 (4) | 3 (7)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 7 (15) | 3 (6) | 2 (9)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (3) | 5 (12) | 2 (2) | 2 (4)
Alanine aminotransferase increased (Investigations) | 1 (2) | 2 (4) | 12 (20) | 5 (6) | 5 (14)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
DOUBLE VISION (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCYTOPENIA (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RBC DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOTAL PROTEIN DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMATOUS RASH TO TRUNK, CHEEKS, EARS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMATUS PRURITIC RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HIVES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERSENSITIFITY & HYPERESETHESIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (9) | 1 (1) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (11) | 3 (7) | 3 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (9) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 1 (2)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 4 (9) | 0 (0) | 3 (9)
Fatigue (General disorders) | 0 (0) | 1 (1) | 5 (7) | 1 (1) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (6) | 1 (1) | 4 (4)
Fever (General disorders) | 0 (0) | 1 (1) | 7 (12) | 2 (2) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 7 (14) | 3 (3) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 9 (12) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 11 (16) | 2 (4) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT03389802/Prot_SAP_000.pdf